CLINICAL TRIAL: NCT00799500
Title: Impact on Prematurity of a First-trimester Screening for Bacterial Vaginosis in Pregnancy Through Weekly Vaginal pH Determination. An Interventional, Community Study.
Brief Title: Bacterial Vaginosis in Pregnancy: Detection by Weekly Vaginal pH Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montse Palacio (Other)
Responsible Party: Sponsor-Investigator, Montse Palacio, MD, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FIS06/0559
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Pregnancy; Bacterial Vaginosis; Preterm Delivery
MeSH Terms: conditions — Vaginosis, Bacterial; Premature Birth | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weekly screening (Experimental): Screening and treatment of bacterial vaginosis during pregnancy through self-administered weekly vaginal pH determination.
  Interventions: Other: Screening
- Observation (No Intervention): Usual care

INTERVENTIONS:
Other: Screening — Weekly vaginal pH
  Arms: Weekly screening

SUMMARY:
Interventional study to assess the effect of early detection and treatment of bacterial vaginosis in pregnancy on preterm delivery rate.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women

Exclusion Criteria:

* Diabetes mellitus (pre-gestational)
* Hypertension (pre-gestational)
* Malformations on ultrasonography at 12 weeks

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Preterm delivery rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Catalonia, Spain